CLINICAL TRIAL: NCT03869840
Title: Accuracy of Detection of Methemoglobin With Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP3186
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Collect Blood Values With Induced Hypoxia, Induced Methemoglobinemia, and Induced Hypoxia and Methemoglobinemia
MeSH Terms: conditions — Methemoglobinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Sensor to spot check blood levels — Sensor to check blood levels, not used as intervention

SUMMARY:
The non-invasive measurement of dysfunctional hemoglobins allows physicians to monitor levels in affected individuals without requiring blood samples or laboratory testing. Nonin Medical Inc, has recently developed a multi-wavelength device that measures carboxyhemoglobin and methemoglobin non-invasively. The primary objective of this study is to validate %MetHb and SpO2 accuracy performance of the study device. Evaluations will be for the range of 0 to 15% MetHb with 95-100% SaO2 as assessed by CO-oximetry, and 0-15% MetHb accuracy under conditions of elevated HHb (SaO2 80-100%) as assessed by CO-oximetry, and SpO2 with 80-100% SaO2 during elevated MetHb as assessed by CO-oximetry.

DETAILED DESCRIPTION:
The goal of this study is to collect data with induced hypoxia, with induced methemoglobinemia, and with induced hypoxia and methemoglobinemia. This will be accomplished in three runs with 24 to 28 plateaus total. The number of plateaus will be dependent on the subject's tolerance of the study procedure. The first run will be strictly induction of hypoxia down to approximately 70% saturation. The second run will be induction of hypoxia down to approximately 80% saturation with mild hypoxia at 7% MetHb. The third run will be induction of hypoxia down to approximately 80% saturation with a target MetHb of 11-15%.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female.
* The subject is of any racial or ethnic group.
* The subject is between 18 years and 50 years of age (self-reported).
* The subject does not have significant medical problems (self-reported).
* The subject is willing to provide written informed consent and is willing and able to comply with study procedures.

Exclusion Criteria:

* Has a BMI greater than 31 (calculated from self-reported weight and height).
* Has had any relevant injury at the sensor location site (self-reported).
* Has a deformity or abnormalities that may prevent proper application of the device under test (based on visual inspection).
* Has a known respiratory condition (self-reported).
* Is currently a smoker (self-reported).
* Has a known heart or cardiovascular condition (self-reported).
* Is currently pregnant (self-reported).
* Is female and actively trying to get pregnant (self-reported).
* Has a clotting disorder (self-reported).
* Has Raynaud's Disease (self-reported).
* Is known to have a hemoglobinopathy such as (anemia, bilirubinemia, sickle-cell anemia, inherited or congenital methemoglobinemia) (self-reported).
* The subject has a COHb greater than 3% or MetHb greater than 2% (based on the first blood sample analysis).
* Has taken blood thinners or medication with aspirin within the last 24 hours (self-reported).
* Has unacceptable collateral circulation from the ulnar artery (based on exam).
* Has donated more than 300 mL of blood within one month prior to start of study (self-reported).
* Is unwilling or unable to provide written informed consent to participate in the study.
* Is unwilling or unable to comply with the study procedures for the primary objectives.
* Has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A minimum of 12 subjects with a minimum of 200 data points for each primary and secondary objective will be enrolled in the study. The subject population will include both male and female subjects and will include a variety of skin tones.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Validate %MetHb | 4 days
  Validate %MetHb accuracy over the range of 0-15% MetHb with SaO2 greater than 95% as assessed by CO-oximetry

SECONDARY OUTCOMES:
Validate the %MetHb accuracy | 4 days
  Validate the %MetHb accuracy with SaO2 greater than 80% as assessed by CO-oximetry An accuracy value (Arms) for %SpO2 over the range of 80-100% SaO2 with elevated MetHb levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States